CLINICAL TRIAL: NCT02643940
Title: The Physiological IMPACT of Coronary Chronic Total Occlusion (CTO) Percutaneous Coronary Intervention (PCI) on Coronary Pressure --Derived Measurements, Its Correlation in the Donor Vessel and the Influence of Collateral Circulation
Brief Title: The Physiological Impact of CTO PCI on Coronary Pressure Measurements and Correlation in Donor Vessel
Acronym: IMPACT-CTO
Status: Completed | Type: Observational
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: B785
Record Dates: First submitted 2015-12-22; First posted 2015-12-31 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Acute Coronary Syndrome; Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention (PCI); Chronic Total Occlusion (CTO); Cardiac MRI; Instantaneous wave-free ratio (iFR)
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (standard care no extra samples collected)
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will be recording pressure wire readings from both blocked and narrowed arteries, to better guide treatment options; medications, stents or potentially bypass surgery, for patients with Chronic Total Occlusion (CTO).

DETAILED DESCRIPTION:
The patients in this study are planned to have a Percutaneous Coronary Intervention (PCI) with recanalization of Chronic Total Occlusion (CTO) on clinical grounds alone.

This study will be recording pressure wire readings from both blocked and narrowed arteries, to better guide treatment option. To date there is no data available on instantaneous wave free ratio (iFR) measurement (a pressure derived assessment of flow limitation) in patients with blocked arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years of age
2. Stable angina / ischaemic symptoms
3. Evidence of viability and / or ischaemia in the chronic total occlusion (CTO) territory
4. Participant is willing and able to give informed consent for participation in the study
5. Presence of a chronic total occlusion (CTO) in RCA:

   * Duration of the occlusion > 3 months;
   * Thrombolysis In Myocardial Infarction (TIMI) (50) coronary flow grade 0;
   * Spontaneously visible collaterals, Rentrop classification grade 1 or 2 or 3 from contralateral donor artery
6. Presence of minor to intermediate coronary stenosis (1-70 %) in the contralateral donor artery
7. Eligible for PCI to a chronic total occlusion (CTO)

Exclusion Criteria:

1. Previous CABG with patent grafts to the interrogated donor artery
2. Left main stenosis of > 40 %
3. Presence of severe flow limiting stenosis in the contralateral donor artery (typically > 70 % stenosis)
4. Haemodynamic instability at the time of intervention (heart rate <40 beats per minute, systolic blood pressure <90mmHg), balloon pump)
5. Significant contraindication to adenosine administration (e.g. heart block, severe asthma)
6. Contraindications to PCI
7. Severe hepatic or lung disease (chronic pulmonary obstructive disease)
8. Pregnancy
9. ACS within 48 hours of procedure
10. Severe valvular heart disease
11. Severe cardiomyopathy / Infiltrative heart disease
12. eGFR < 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for a PCI CTO
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Coronary pressure changes | 5 Minutes
  Changes in coronary pressure - derived measurements (resting Pd/Pa, iFR and FFR) in donor artery pre and post RCA CTO PCI

SECONDARY OUTCOMES:
Population correlation | 5 minutes
  Correlation between coronary pressure---derived measurements in this population.
Donor artery correlation | 5 minutes
  Correlation between collateral circulation function on coronary pressure - derived measurements in donor artery pre and post RCA CTO PCI.
Cardiac MRI correlation | 5 minutes
  Correlation between baseline coronary pressure - derived measurements in donor artery pre RCA CTO PCI, collateral circulation indices and baseline non-invasive functional assessment /Cardiac MRI (CMR)
Effects of stenosis severity (QCA) | 5 minutes
  Effects of stenosis severity (QCA) in donor artery on coronary pressure-derived measurements
Collateral circulation characteristics | 5 minutes
  Influence of collateral circulation characteristics on coronary pressure-derived measurements
Coronary pressure and jeopardy scores correlation | 5 minutes
  Correlation between coronary pressure-derived measurements in the donor artery and myocardial jeopardy scores in the donor artery

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Keeble, MBBS MRCP, Principal Investigator — The Essex Cardiothoracic Centre
Locations (1):
- The Essex Cardiothoracic Centre, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Karamasis GV, Kalogeropoulos AS, Mohdnazri SR, Al-Janabi F, Jones R, Jagathesan R, Aggarwal RK, Clesham GJ, Tang KH, Kelly PA, Davies JR, Werner GS, Keeble TR. Serial Fractional Flow Reserve Measurements Post Coronary Chronic Total Occlusion Percutaneous Coronary Intervention. Circ Cardiovasc Interv. 2018 Nov;11(11):e006941. doi: 10.1161/CIRCINTERVENTIONS.118.006941. PMID 30571203
- [Result] Mohdnazri SR, Karamasis GV, Al-Janabi F, Cook CM, Hampton-Till J, Zhang J, Al-Lamee R, Dungu JN, Gedela S, Tang KH, Kelly PA, Davies JE, Davies JR, Keeble TR. The impact of coronary chronic total occlusion percutaneous coronary intervention upon donor vessel fractional flow reserve and instantaneous wave-free ratio: Implications for physiology-guided PCI in patients with CTO. Catheter Cardiovasc Interv. 2018 Sep 1;92(3):E139-E148. doi: 10.1002/ccd.27587. Epub 2018 Mar 22. PMID 29569332